CLINICAL TRIAL: NCT03518346
Title: Use of Virtual Reality Game Playing During Venipuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1170355
Record Dates: First submitted 2018-03-27; First posted 2018-05-08 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Autism; Development Delay; Typical Development
MeSH Terms: conditions — Autistic Disorder; Learning Disabilities | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Participants may be randomized to the virtual reality, VR, group or the standard of care group. For the VR group, we are using the Samsung VR Go (VR head set), Samsung S7 (phone) and programmed distraction (Spaceburgers, Pebbles the Penguin, and/or Happy Place). Spaceburgers and Pebbles the Penguin were designed by the Department of Anesthesiology at Lucile Packard Children's Hospital Stanford through the Stanford Chariot Program (Childhood Anxiety Reduction Through Innovation and Technology). Happy Place is a nongame immersive experience that will be offered to children uninterested in the previously mentioned game. Happy Place was designed by a Swedish Pharmacy Chain, Apotek Hjartat, aimed to distract patients from their pain with a peaceful, interactive environment. Each of the video games runs for the length of time needed to complete the venipuncture.
  Interventions: Behavioral: Virtual Reality
- Standard of Care Group (Active Comparator): Participants may be randomized to the virtual reality, VR, group or the standard of care group. The standard of care group will use various distractions. Distraction tools include books and movies using a wall mounted TV as standard practice.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Virtual Reality — Samsung VR Go (VR head set), Samsung S7 (phone), and programmed distraction
  Arms: Virtual Reality Group
Behavioral: Standard of Care — Books, movies, TV
  Arms: Standard of Care Group

SUMMARY:
To evaluate the impact of using virtual reality, VR, game playing on successful completion and reduction of distress and pain in pediatric venipuncture, and to increase adherence in obtaining the desired blood volume.

DETAILED DESCRIPTION:
Participants will be randomly assigned using a random number generator to either the virtual reality condition, or to the standard procedure that includes using books and/or watching movies as a standard method of distraction.

Participants will take part in the study during their scheduled research venipuncture. The venipuncture lasts approximately 15-30 minutes. Pre and post venipuncture questionnaires for both participant and parent will take 15 minutes to complete. Total study time is between 30 and 45 minutes. Questionnaires completed by research personal will take 15 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 8-19 years old that are receiving a blood draw as part of their ReCHARGE evaluation
2. History of distress or refusal of blood draws or similar medical procedures OR
3. Parent or child endorsement of fear, anxiety, concern or adherence in past blood draw during the recruitment phone call, consent or child evaluation will be offered the potential of the VR intervention OR
4. Endorsement of anxiety or concerns with medical procedures on an in house phlebotomist blood draw screening form will also be used as inclusion criteria.

Exclusion Criteria:

1. History of seizures.
2. Vision loss or significant visual impairment to the degree that the participant is unable to see the activity and features of the VR game.

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Attempting vs. Refusing Venipuncture | 2 years
  Compare if the participant is willing to let us attempt the venipuncture or refuses the venipuncture. the number of patients will be counted.

SECONDARY OUTCOMES:
Blood volume | 2 years. Collected once on each participant: immediately following injection
  Volume of blood collected in mL
Pain Scale | 2 years. Collected once on each participant: immediately following injection
  Pain scale measures patient reports of pain levels after venipuncture on scale of 0-10
Satisfaction Survey | 2 years. Collected once on each participant: immediately following injection
  Child and Parent Satisfaction Survey consists of 5 questions with likert scale responses
Fear Scale | 2 years. Collected twice on each participant: before and immediately following injection
  Child Fear scale measures patient reports of fear levels before and after venipuncture on scale of 0-4
Time to Achieve Optimal Blood Volume | 2 years. Collected on each participant: during venipuncture procedure
  Time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Julie Schweitzer, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis MIND Institute, Sacramento, California, United States